CLINICAL TRIAL: NCT03777462
Title: Comparisons of Different Neoadjuvant Chemotherapy Regimens With or Without Stereotactic Body Radiation Therapy for Borderline Resectable Pancreatic Cancer: Study Protocol of a Prospective, Randomized Phase II Trial
Brief Title: Borderline Resectable Pancreatic Cancer Neoadjuvant Chemoradiotherapy Clinicaltrial-1
Acronym: BRPCNCC-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Research assistant of Hepatobiliary and Pancreatic Surgery, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP04
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; neoadjuvant chemotherapy; SBRT
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A of neoadjuvant chemotherapy (Active Comparator): Neoadjuvant gemcitabine plus nab-paclitaxel is used in this group. Intravenous administration of gemcitabine (1000mg/m2) and nab-paclitaxel (125 mg/m2) are initiated on day 1, 8 and 15 during each 4-week cycle, which will repeat for 3 cycles. And surgical resection is performed after completion of the whole chemotherapy.
  Interventions: Drug: Neoadjuvant gemcitabine plus nab-paclitaxel
- Group B of neoadjuvant chemoradiotherapy (Experimental): Neoadjuvant gemcitabine plus nab-paclitaxel with SBRT is used in this group. Intravenous administration of gemcitabine (1000mg/m2) and nab-paclitaxel (125 mg/m2) are initiated on day 1, 8 and 15 during each 4-week cycle, which will repeat for 3 cycles. After completion of the whole chemotherapy, patients will first receive PET-CT to exclude distant metastases and then undergo SBRT. The prescribed dose is 7.5-8Gy/f for 5 fractions. Dose constraints of normal tissues are referred to the American Association of Physicists in Medicine guidelines in TG-101. And surgical resection is performed 3 weeks after SBRT.
  Interventions: Drug: Neoadjuvant gemcitabine plus nab-paclitaxel with SBRT
- Group C of neoadjuvant chemoradiotherapy (Experimental): Neoadjuvant S-1 plus nab-paclitaxel with SBRT is used in this group. Intravenous administration of nab-paclitaxel (125 mg/m2) is initiated on day 1, 8 and 15 during each 4-week cycle, which will repeat for 3 cycles. And S-1 is orally administrated at a dose of 80 mg/m2 for 18 days followed by a 10-day rest during each 4-week cycle, which aslo continues for 3 cycles. After completion of the whole chemotherapy, patients will first receive PET-CT to exclude distant metastases and then undergo SBRT. The prescribed dose is 7.5-8Gy/f for 5 fractions. Dose constraints of normal tissues are referred to the American Association of Physicists in Medicine guidelines in TG-101. And surgical resection is performed 3 weeks after SBRT.
  Interventions: Drug: Neoadjuvant S-1 plus nab-paclitaxel with SBRT

INTERVENTIONS:
Drug: Neoadjuvant gemcitabine plus nab-paclitaxel — Neoadjuvant gemcitabine plus nab-paclitaxel is used in the intervention group for 3 cycles. Standard doses of gemcitabine and nab-paclitaxel are adopted. Surgical resection will be performed after neoadjuvant chemotherapy.
  Arms: Group A of neoadjuvant chemotherapy
Drug: Neoadjuvant gemcitabine plus nab-paclitaxel with SBRT — Neoadjuvant gemcitabine plus nab-paclitaxel with SBRT is used in the intervention group for 3 cycles. Standard doses of gemcitabine and nab-paclitaxel are adopted. The radiation dose of SBRT is 7.5-8Gy/f for 5 fractions. Surgical resection will be performed 3 weeks after SBRT.
  Arms: Group B of neoadjuvant chemoradiotherapy
Drug: Neoadjuvant S-1 plus nab-paclitaxel with SBRT — Neoadjuvant S-1 plus nab-paclitaxel with SBRT is used in the intervention group for 3 cycles. Standard doses of gemcitabine and nab-paclitaxel are adopted. The radiation dose of SBRT is 7.5-8Gy/f for 5 fractions. Surgical resection will be performed 3 weeks after SBRT.
  Arms: Group C of neoadjuvant chemoradiotherapy

SUMMARY:
This study is to investigate whether neoadjuvant chemotherapy plus SBRT results in better outcomes compared with neoadjuvant chemotherapy alone and also compare the efficacy of gemcitabine plus nab-paclitaxel with SBRT and S-1 plus nab-paclitaxel with SBRT.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial that investigate whether neoadjuvant chemotherapy plus SBRT results in better outcomes compared with neoadjuvant chemotherapy alone and also compare the efficacy of gemcitabine plus nab-paclitaxel with SBRT and S-1 plus nab-paclitaxel with SBRT. It is known that neoadjuvant therapy is vital for improved survival, which has been confirmed in previous studies that neoadjuvant chemotherapy with or without radiotherapy provides superior overall compared with upfront surgery. However, question of whether the addition of radiotherapy to neoadjuvant chemotherapy can improve prognosis compared with chemotherapy alone is a challenging matter. Also, no studies have evaluated the efficacy of S-1 as the neoadjuvant chemotherapy regimen for BRPC albeit similar prognosis has been found between S-1 and gemcitabine in advanced pancreatic cancer. In this trial, patients with biopsy and radiographically confirmed BRPC will be randomly allocated into three groups: neoadjuvant gemcitabine plus nab-paclitaxel, neoadjuvant gemcitabine plus nab-paclitaxel with SBRT and neoadjuvant S-1 plus nab-paclitaxel with SBRT. Surgical resection will be performed 3 weeks after SBRT. The primary endpoint is overall survival. The secondary outcomes are progression free survival, pathological complete response rate, R0 resection rate and incidence of adverse effects. If results show the survival benefits of neoadjuvant chemotherapy plus SBRT and similar outcomes between S-1 and gemcitabine, it may provide evidence of clinical practice of this modality for BRPC.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old and ≤80 years old;
* Histological proven pancreatic adenocarcinoma;
* Borderline resectable pancreatic cancer proven by imaging examinations via multidisciplinary approaches according to NCCN guidelines;
* No prior chemotherapy or radiotherapy;
* ECOG of 0 or 1;
* Routine blood test: absolute neutrophil count>1500/mm3, platelet>100000/mm3;
* Normal liver function: serum total bilirubin≤2.0mg/dl, ALT and AST<2.5 times of the upper limit of normal value;
* Normal kidney function: serum creatinine<1.5 times of the upper limit of normal value or creatinine clearance rate>45ml/min;
* No severe comorbidities.

Exclusion Criteria:

* Metastatic pancreatic cancer;
* Patients who had surgeries, chemotherapy or other treatments before inclusion;
* Impaired organ functions: heart failure (New York Heart Association III-IV), coronary heart disease, myocardial infarction within 6 months, severe cardiac arrhythmia and respiratory failure;
* Confirmed other cancer within 5 years;
* Pregnant women or lactating women;
* Patients enrolled in other clinical trials or incompliant of regular follow up;
* Patients who did not provide an informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall time | From date of randomization until the date of death from any cause, whichever came first, assessed up to 24 months
  The time between operation and the death of patients

SECONDARY OUTCOMES:
Disease free time | From date of randomization until the date of first documented progression or metastasis, assessed up to 12 months
  The time between operation and the relapse or metastasis of tumors

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, Doctor, Principal Investigator — Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Gao S, Zhu X, Shi X, Cao K, Bian Y, Jiang H, Wang K, Guo S, Zhang H, Jin G. Comparisons of different neoadjuvant chemotherapy regimens with or without stereotactic body radiation therapy for borderline resectable pancreatic cancer: study protocol of a prospective, randomized phase II trial (BRPCNCC-1). Radiat Oncol. 2019 Mar 27;14(1):52. doi: 10.1186/s13014-019-1254-8. PMID 30917842